CLINICAL TRIAL: NCT02209961
Title: To Check the Efficacy and Saftey of Combined Ex-PRESS Implantation Alone or With Phacoemulsification for Glaucoma Associated With Cataract
Brief Title: Combined Ex-PRESS Implantation Alone or With Phacoemulsification for Glaucoma Associated With Cataract
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0054-13
Record Dates: First submitted 2014-03-19; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- glaucoma and ocular hypertension: glaucoma and ocular hypertension

SUMMARY:
A prospective study reporting on Ex-PRESS shunt implantation alone or combined cataract and glaucoma surgery.

DETAILED DESCRIPTION:
The occurrence of both glaucoma and clinically relevant cataract in the same individual is a frequent condition, especially in the elderly population. Besides age, this might be related to the possible role of antiglaucoma medications in the progression of lens opacity.When both procedures are required, these can be performed separately or in combination.

Glaucoma filtering surgery is indicated when glaucomatous damage progresses despite the lower level of intraocular pressure (IOP) obtained with pharmacological and/or laser treatment.

The Ex-PRESS is a miniature stainless steel glaucoma device, developed as an alternative to trabeculectomy and to the other types of glaucoma filtering surgery for patients with POAG. This procedure would be theoretically more reproducible and simple to perform as well as less traumatic to the ocular tissue than traditional filtering surgery. The implant is inserted at the limbus under a conjunctival flap and diverts the aqueous humour from the anterior chamber to the subconjunctival space, obtaining the formation of a conjunctival filtration bleb, in a similar way to trabeculectomy. This procedure can be performed on its own or in combination with phacoemulsification.

This study is aimed to test the efficacy and saftey of Ex-PRESS shunt implantation alone or combined cataract and glaucoma surgery in patients with medically uncontrolled glaucoma and cataract .

ELIGIBILITY:
Inclusion Criteria:

- age above 18

Exclusion Criteria:

- congenital glaucoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with uncontrolled glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure change in Ex-PRESS shunt implantation alone or combined cataract and glaucoma surgery in patients with medically uncontrolled glaucoma and cataract . | within one to two years post surgery
  to check the change in intraocular pressure after EX-PRESS shunt implantation

CONTACTS AND LOCATIONS:
Overall Officials: Rana N Hanna, M.D, Principal Investigator — Hillel Yaffe Medical Center